CLINICAL TRIAL: NCT01675700
Title: Topical Nitrates for Myofascial Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GF Strong Rehabilitation Centre (Other)
Responsible Party: Principal Investigator, Anibal Bohorquez, Medical Resident, GF Strong Rehabilitation Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 122975
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Myofascial Trigger Points
Keywords: Myofascial pain; Trigger point; Nitroglycerin
MeSH Terms: interventions — Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Myofascial trigger point (Experimental): Patients diagnosed with myofascial trigger points who will receive a nitroglycerin patch over the trigger point.
  Interventions: Drug: Nitroglycerin patch

INTERVENTIONS:
Drug: Nitroglycerin patch — Nitroglycerin 0.1 mg/hr patch
  Other Names: Nitro-Dur 0.1

SUMMARY:
The purpose of this study is to determine whether a topical nitroglycerine patch applied daily over a trapezius trigger point can improve patients' symptoms.

If there is improvement, this open label study will help determine the degree of improvement and contribute to the design of a larger double blind placebo controlled trial.

We would consider moving forward to a large randomized trial if:

* The intervention is acceptable to patients (>= 70%) and
* Compliance is satisfactory (>=80%) and
* We find preliminary evidence of efficacy, i.e. average reduction in pain of 20mm on the VAS.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include age between 19 and 65 years old, myofascial pain lasting at least 6 months, and a myofascial trigger point point in the trapezius muscle.

Exclusion Criteria:

* Our exclusion criteria include symptomatic disc herniation, symptomatic cervical osteoarthritis, systemic infection, malignancy, collapsed vertebra, thoracic outlet syndrome, temporomandibular joint dysfunction, collagen-vascular disease, or brachial plexopathy. Patients with ongoing litigation regarding their symptoms are not eligible for this study. Also excluded are patients with underlying cardiac disease, hypotension, or medical conditions that may not allow them to tolerate the use of vasodilators, and those who use phosphodiesterase inhibitors.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Pain at the time of clinic visit and over the previous week as measured by a Visual Analog Scale, VAS, for pain and a pressure algometer measurement to obtain pressure pain thresholds over the patients trigger point. | 1 month

SECONDARY OUTCOMES:
As another secondary outcome we will ask the participants whether the benefits of the treatment are good enough that they would continue using the nitroglycerin patch. This will be a yes or no response. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Hubert A Anton, MD, Principal Investigator — University of British Columbia